CLINICAL TRIAL: NCT02513095
Title: Phase 2, Single-Site, Open-Label, Randomized, 2-Arm Parallel Study to Assess the Efficacy and Safety of Ryanodex® (EGL-4104) as Adjuvant Treatment in Subjects With Exertional Heat Stroke (EHS)
Brief Title: Efficacy and Safety of Ryanodex® (EGL-4104) as Adjuvant Treatment in Subjects With Exertional Heat Stroke (EHS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eagle Pharmaceuticals, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGL-4104-C-1502
Record Dates: First submitted 2015-07-21; First posted 2015-07-31 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Heat Stroke
MeSH Terms: conditions — Heat Stroke | interventions — Dantrolene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ryanodex (Experimental): Ryanodex (dantrolene sodium) for injectable suspension administered as an IV bolus, in addition to standard of care (SOC) treatment.
  Interventions: Drug: Dantrolene sodium for injectable suspension
- Standard of Care only (SOC) (No Intervention): Standard of Care (SOC) treatment only, consisting of body cooling and supportive measures implemented immediately.

INTERVENTIONS:
Drug: Dantrolene sodium for injectable suspension — Ryanodex will be administered as a rapid IV push as a single doses of 2 mg/kg or as 1 mg/kg.
  Other Names: Ryanodex; EGL-4104
  Arms: Ryanodex

SUMMARY:
Study EGL-4104-C-1502 is a phase 2, single-site, open-label, randomized, 2-arm parallel study of Ryanodex for the adjuvant treatment of exertional heat stroke (EHS) administered intravenously (IV), to current standard of care (SOC). SOC for the treatment of EHS is defined as effective body cooling, which should be implemented as quickly as available after diagnosis of exertional heat stroke.

DETAILED DESCRIPTION:
The study will take place at emergency medical facilities.

Due to the life-threatening nature of exertional heat stroke (EHS), rapid assessment for inclusion into the study and subsequent immediate treatment must occur. Following initial triage and primary assessment of a subject, the subject's baseline status should be documented, and once a diagnosis of EHS is obtained, SOC treatment will be initiated immediately, the subject will be randomized to one of two treatment arms (SOC only or SOC plus Ryanodex).

Patients will be remain hospitalized for up to 72 hours after administration of the first dose of study drug and implemented SOC and will receive all necessary supportive measures until resolution of symptoms.

Study duration: 72 hours

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be entered in the study if they have a core body temperature obtained rectally of ≥ 40.0°C (104°F)
* Recent history or suspected recent history (prior 24 hours) of performing intense physical activity (exertional activity)
* The subject has an impaired consciousness level as evidenced by a GCS score < 13
* The subject has tachycardia (heart rate ≥ 100 bpm)

Exclusion Criteria:

* The subject is diagnosed with or is suspected of having an acute clinically severe infection, which in the opinion of the Investigator may increase the subject's risk for participating in the study and/or may impair the ability of performing and/or interpreting study assessments
* The subject has severe hyperthermia secondary to a condition other than heat stroke (e.g., serotonin syndrome, thyrotoxicosis, pheochromocytoma, or brain hemorrhage)
* There is likelihood of head trauma in the past 6 months, or other significant cardiovascular, pulmonary, hepatic, endocrine, or renal illness that in the opinion of the Investigator may increase the subject's risk for participating in the study and/or may impair the ability of performing and/or interpreting study assessments
* A female subject has a positive pregnancy test (urine) or evidence of active lactation
* Reported known use of potent CYP3A4 inhibitors
* A known history of allergy or hypersensitivity to dantrolene
* A history of chronic and ongoing assisted mechanical ventilation prior to the onset of EHS via an established artificial or supported airway (e.g., for severe chronic obstructive pulmonary disease [COPD], upper airway disease, impaired respiratory function). Note: Endotracheal intubation and mechanical ventilation as part of supportive measures for the treatment of EHS are allowed

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hepner, MD, Study Director — Eagle Pharmaceuticals, Inc.
Locations (1):
- Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to the life-threatening nature of EHS, eligible subjects were immediately randomized to enter the study Treatment Phase (up to 120 minutes duration)
Groups:
- Active: Ryanodex plus Standard of Care
- Control: Standard of Care Only
Period: Overall Study
Arm/Group | Active | Control
Started | 17 | 17
Treatment Phase - Up to 120 Minutes | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ryanodex Plus Standard of Care: Ryanodex (dantrolene sodium) for injectable suspension administered as an IV bolus, in addition to standard of care (SOC) treatment.
  Dantrolene sodium for injectable suspension: Ryanodex will be administered as a rapid IV push as a single doses of 2 mg/kg or as 1 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Ryanodex Plus Standard of Care | Standard of Care Only (SOC) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 1 | 2 | 3
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Glasgow Coma Scale [Mean (Standard Deviation); unit: units on a scale] — Cumulative incidence of subjects achieving a Glasgow Coma Scale(GCS) ≥ 13 at or prior to 90 minutes post-randomization. The Glasgow Coma Scale (GCS) is a reliable and objective way of recording the initial and subsequent level of consciousness in a person after a brain injury. The range of total GCS score is 3 to15 where a higher GCS score represents a better outcome. The scores of subscales are summed to determine the total score. A GCS score of 13-15 is considered Mild; a GCS score of 9-12 is considered Moderate; and a GCS score of 3-8 is considered Severe.
  units on a scale | 6.1 (3.98) | 5.9 (3.18) | 6.0 (3.55)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Recovery of Level of Consciousness Defined as a Glasgow Coma Scale (GCS) GCS ≥ 13
Description: Number of subjects achieving a Glasgow Coma Scale(GCS) ≥ 13 at or prior to 90 minutes post-randomization. The Glasgow Coma Scale (GCS) is a reliable and objective way of recording the initial and subsequent level of consciousness in a person after a brain injury. The range of total GCS score is 3 to15 where a higher GCS score represents a better outcome. The scores of subscales are summed to determine the total score*. A GCS score of 13-15 is considered Mild impairment of consciousness; a GCS score of 9-12 is considered Moderate impairment of consciousness; and a GCS score of 3-8 is considered Severe.
  *Subscales: Eyes Response -Spontaneous=4; To sound =3; To Pressure=2; None=1; not tested. Verbal Response- Oriented=5; Confused=4; Words=3; Sounds=2; None-1; Not tested. Motor Response: Obeys Commands=6; Localizes=5; Normal Flexion=4; Abnormal Flexion=3; Extension=2; None=1; Not tested.
Time Frame: 90 minutes post-randomization
Measure: Count of Participants; unit: Participants
Groups:
- Ryanodex Plus Standard of Care: Ryanodex plus Standard of Care. Ryanodex will be administered as a rapid IV push as a single doses of 2 mg/kg or as 1 mg/kg.
- Standard of Care: Standard of Care Only
Arm/Group | Ryanodex Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 17 | 17
Participants | 5 | 2
Statistical Analysis 1: Comparison: Ryanodex Plus Standard of Care vs Standard of Care; Test type: Superiority; p = 0.396, Chi-squared, Corrected; Odds Ratio (OR) = 6, 95% CI 2-sided [0.6 to 76.8]

ADVERSE EVENTS:
Time Frame: .Up to 30 days post-discharge.
Arm/Group | Ryanodex | Standard of Care Only (SOC)
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 4/17 | 3/17
Other Adverse Events (participants affected / at risk) | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ryanodex (N=17) | Standard of Care Only (SOC) (N=17)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ryanodex (N=17) | Standard of Care Only (SOC) (N=17)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 2 (2) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 2 (2)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Investigations) | 2 (2) | 0 (0)
Hypoglycemia (Investigations) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 3 (3)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI has no right to discuss/publish/disclose the trial data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol Synopsis (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT02513095/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistics (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT02513095/SAP_001.pdf